CLINICAL TRIAL: NCT05215080
Title: The Tolerance of Organic Formula Milk and Its Fecal Microbiome Characteristic in Infants
Acronym: TOFeM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Collaborators: Arla Foods (Industry)
Responsible Party: Principal Investigator, Bahrul Fikri, Medical doctor, Doctor of Philosophy, Principal Investigator, Hasanuddin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRP/2021/XI/001/AFA
Record Dates: First submitted 2021-12-08; First posted 2022-01-31 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Food Allergy in Infants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Group of infants aged 6-7 months that given organic formula milk three times a day for three months. Each serving contains 7 spoons (1 spoon contain 4,6 grams) of milk powder and 210 ml of water.
  Interventions: Dietary Supplement: Organic Formula Milk

INTERVENTIONS:
Dietary Supplement: Organic Formula Milk — Organic formula milk is given to the infants three times a day for three months. Each serving contains 7 spoons (1 spoon contain 4,6 grams) of milk powder and 210 ml of water.

SUMMARY:
This interventional study aims to investigate the tolerance of organic formula milk on infants supplemented with organic formula milk. This study also observes gut microbiota, short chain fatty acids, nutritional status, and atopic manifestation on infants supplemented with organic formula milk. This study will be done on 50 subjects, with an age of 6-7 months old, 38-42 weeks of gestation, had a birth weight ranging from 2700 grams to 4200 grams, not suffering from any major congenital anomaly, not severely stunted at birth, has a normal thyroid function, not suffering any prominent gastrointestinal disease, not having a severe disease at the beginning of study, and has an approval from their parents. Participants' diet will be added an organic formula for infant for 3 months, and will be monitored regularly, since this study starts, at each month, and at the end of this study. The participants' gut microbiomes will be calculated at every session of monitoring by collecting their fecal samples, and brought to laboratory. Anthropological data (weight, height, body mass index), atopic manifestation, IL-6 and IL-10 will also be collected.

DETAILED DESCRIPTION:
All the guardians or parents of the participants in this study will be interviewed in order to record the dietary and sign for inform consent. Parents will be given a journal to record the participant's diet, any sign of colic on subjects, quality of sleep, and wellbeing. All the participants will be fed organic formula milk as a part of their dietary for 12 weeks. Before feeding the formula, the nutritional status will be measured and the participant's fecal will be collected for microbiome and short chain fatty acid (SCFA) examination. Every month the parents will be called in order to assess for child's sickness, allergy, body weight, length, head circumference, and to review their journal.

A visit follow up will be done before and after the study, the tolerance, nutritional status (including body mass index) and fecal collection for all subjects will be performed. The investigators will also collect the allergy related data. Each fecal examination will follow a strict cold chain procedure, each sample will be collected directly, bottled, and frozen to minimize error. The frozen samples will be transported in insulated bags with frozen ice blocks before being transferred to -80°C for storage.

A statistical analysis will be performed using r program and STATA 13.0. The Normality of data distribution will be tested using the Shapiro-Wilk test. To evaluate potential associations between factors in relation to fecal microbiome or SCFAs, Spearman's rank correlations will be calculated. A p-value <0.05 will be considered significant.

The model will be adjusted for potential confounders. Estimated associations will be described as odds ratios (ORs) with 95% confidence intervals (CIs). The non-parametric Wilcoxon test for paired samples will be used to compare different laboratory parameters at different times of collecting samples. The Mann-Whitney U test for unpaired samples will be applied to compare different categorical parameter between infants before and after treatment. Multivariable linear regressions will be done to find out the association of different parameters change before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 6-7 months of age.
* Gestational age 38-42 weeks
* Birth weight >2700 and <4200 gram
* Not suffering from a major congenital anomaly, severely stunted at birth, not having a thyroid problem, not suffered from prominent gastrointestinal diseases, severe diseases at the time of inclusion (severe pneumonia, severe dehydration, etc)
* Parents want to follow the study by signing the informed consent

Exclusion Criteria:

* Subjects are in the severe disease condition at the time of recruitment
* Severe acute malnutrition
* Have conditions that will influence the nutritional status such as moderate to severe dehydration, organomegaly, edema.

Ages: 6 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Participants with diarrhea defined by WHO definition of diarrhea | 12 weeks
  Evaluate the acceptability of organic formula milk on infants by observing the stool consistency and frequency of passing stool
Participants with atopic dermatitis in Hanifin-Rajka criteria | 12 Weeks
  Evaluate any atopic dermatitis manifestation arise during organic formula milk consumption based on Hanifin Rajka Criteria
Participants with food allergy measured by positive Oral Food Challenge | 12 Weeks
  Evaluate any allergic reaction during organic formula milk consumption based on positive oral food challenge

SECONDARY OUTCOMES:
Diversity of gut microbiota in operational taxonomic unit | 12 weeks
  Fecal samples obtained and fresh frozen by liquid nitrogen for 16S rRNA analysis Genomic DNA was extracted from fecal samples and purified using Genomic DNA from stool samples (Macherey-Nagel GmbH & Co. KG, Germany). Each DNA specimen from feces was amplified using the Ion 16S Metagenomics Kit (Thermo Fisher Scientific, Bremen, Germany). The amplicons were purified and prepared for the sequencing library by using the Ion Plus Fragment Library Kit (Thermo Fisher Scientific) and the Ion Personal Genome Machine (PGM) Hi-Q sequencing kit following the protocol of the kit. The sequencing runs were performed on the Ion PGM platform (Thermo).
Abundance of gut microbiota in operational taxonomic unit | 12 weeks
  Fecal samples obtained and fresh frozen by liquid nitrogen for 16S rRNA analysis Genomic DNA was extracted from fecal samples and purified using Genomic DNA from stool samples (Macherey-Nagel GmbH & Co. KG, Germany). Each DNA specimen from feces was amplified using the Ion 16S Metagenomics Kit (Thermo Fisher Scientific, Bremen, Germany). The amplicons were purified and prepared for the sequencing library by using the Ion Plus Fragment Library Kit (Thermo Fisher Scientific) and the Ion Personal Genome Machine (PGM) Hi-Q sequencing kit following the protocol of the kit. The sequencing runs were performed on the Ion PGM platform (Thermo).
Concentration of gut short chain fatty acids in mMol | 12 weeks
  Faecal samples obtained. Reagen used is N-tert-butyldimethylsilyl-N-trifluoroace- tamide (MTBSTFA) (Sigma-Aldrich, St. Louis, MO, USA) and analysis was performed using gas chromatogra- phy-tandem mass spectrometry (GC/MS/MS) platforms on a Shimadzu GCMS-TQ8030 triple quadrupole mass spectrometer (Shimadzu, Kyoto, Japan) with a capillary column (BPX5) (SGE Analytical Science Pty. Ltd., Melbourne, Australia).
Body weight in kilograms measured with Krisbow electronic baby scale 10110689 | 12 weeks
  Measurements of weight every 4 weeks
Body length in centimeters measured with Krisbow electronic baby scale 10110689 | 12 weeks
  Measurements of length every 4 weeks
Head circumference measured with Onemed medline tape measure | 12 weeks
  Measurements of head circumference every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bahrul Fikri, MD, PhD, Principal Investigator — Hasanuddin University
Locations (1):
- Hasanuddin University, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
We are going to share individual participant data that underlie results in this publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: The data will be shared by email sent by the primary investigator

REFERENCES:
- [Background] Ohno H. Gut microbial short-chain fatty acids in host defense and immune regulation. Inflammation and regeneration. 2015;35:114-121
- [Background] Inoue Y, Shimojo N. Microbiome/microbiota and allergies. Semin Immunopathol. 2015 Jan;37(1):57-64. doi: 10.1007/s00281-014-0453-5. Epub 2014 Oct 18. PMID 25326106
- [Background] Sakurai K, Miyaso H, Eguchi A, Matsuno Y, Yamamoto M, Todaka E, Fukuoka H, Hata A, Mori C; Chiba study of Mother and Children's Health Group. Chiba study of Mother and Children's Health (C-MACH): cohort study with omics analyses. BMJ Open. 2016 Jan 29;6(1):e010531. doi: 10.1136/bmjopen-2015-010531. PMID 26826157
- [Background] Simonyte Sjodin K, Vidman L, Ryden P, West CE. Emerging evidence of the role of gut microbiota in the development of allergic diseases. Curr Opin Allergy Clin Immunol. 2016 Aug;16(4):390-5. doi: 10.1097/ACI.0000000000000277. PMID 27253486

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT05215080/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT05215080/ICF_001.pdf